CLINICAL TRIAL: NCT01333150
Title: Effects of a Low-dose Propranolol on a Stress Induced Autonomic Response and on Muscle Pain
Brief Title: Effect of Propranolol on the Autonomic Nervous System and Muscle Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: M-20090062
Record Dates: First submitted 2011-03-30; First posted 2011-04-11 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Temporomandibular Joint Disorders; Myofascial Temporomandibular Disorders
Keywords: Temporomandibular disorders; Orofacial pain
MeSH Terms: conditions — Temporomandibular Joint Disorders; Facial Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propranolol (Experimental)
  Interventions: Drug: Propranololhydrochlorid
- Placebo (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propranololhydrochlorid — One single dose of Propranolol tablet of 40 mg randomized in one of the two sessions
  Other Names: Propranolol "DAK" 40 mg, Nycomed Denmark ApS
  Arms: Propranolol
Drug: Placebo — One single dose of placebo
  Arms: Placebo

SUMMARY:
The project's primary purpose is to test the hypothesis that oral administration of a low single dose of β-antagonist propranolol (40 mg) reduces pain sensitivity in patients with masticatory muscle pain.

ELIGIBILITY:
Inclusion Criteria:

* Meet Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD) for myofascial TMD diagnosis corresponding to group 1a or 1b
* Characteristic Pain Intensity (CPI) more than or equal to 20 (Axe II, RDC/TMD questionnaire)
* Women of childbearing potential must use adequate contraception
* Signed consent statement

Exclusion Criteria:

* Other acute pain cause such as acute toothache or a pain condition the investigator estimates to be contraindicated for participation in the experiment
* Recognized existing malignancy or within last 5 years
* Known HIV
* Abuse of drugs including alcohol
* Recognized Raynaud's syndrome
* Former sympathectomy
* Known cardiovascular disease including abnormal EKG and blood pressure (ECG-12 is recorded before the first trial session and assessed by the physician)
* Recognized lung insufficience, including bronchial asthma
* Known severe hepatic or renal dysfunction
* Known diabetes mellitus
* Known severe depression
* Pregnancy (tests performed in both sessions 1 and 2 before the start of a session)
* Fertility Treatment
* Lactation
* Post-menopausal
* Previous adverse reaction when taking beta-blocker, including hypersensitivity to propranolol or to any of the excipients
* Patients who can not read and understand the written information
* Patients who can not follow the protocol
* Patients who do not agree to comply with the requirements for participation in both studies regarding food intake, physical activity, etc.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Participants will be asked to score their actual pain level in both of the two experimental sessions they will participate in; an expected average of two weeks between the two sessions
  Numeric Rating Scale 0-10

SECONDARY OUTCOMES:
Haemodynamic parameters | Participants will be monitored during the entire session in both of the two experimental sessions they will participate in; an expected average of two weeks between the two sessions
  Monitoring of pulse and blodpressurevariability, respiration, baroreceptor sensitivity, measured non-invasively by Task Force Monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Svensson, DDS, PhD, Dr.Odont, Principal Investigator — University of Aarhus
Locations (2):
- Denmark (2):
  - Section of Clinical Oral Physiology,Department of Dentistry,HEALTH. Aarhus University, Aarhus
  - Section of Clinical Oral Physiology, Aarhus University, Aarhus C